CLINICAL TRIAL: NCT00742209
Title: Study MPX111381: A Dose-ranging Study Evaluating the Efficacy, Safety and Tolerability of GSK1838262 (XP13512) in the Prophylactic Treatment of Migraine Headache
Brief Title: Prevention Study in Adult Patients Suffering From Migraine Headaches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 111381
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Results first posted 2011-12-05 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2011-10

CONDITIONS: Migraine Disorders; Migraine
Keywords: migraine; prophylaxis; prevention
MeSH Terms: conditions — Migraine Disorders | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): PBO
  Interventions: Drug: Placebo
- GSK 1838262 1200 mg/day (Active Comparator): 600 or 1200 mg/day
  Interventions: Drug: GSK1838262
- GSK 1838262 1800 mg/day (Active Comparator): 600 or 1200 or 1800 mg/day
  Interventions: Drug: GSK1838262
- GSK 1838262 2400 mg/day (Active Comparator): 600 or 1200 or 1800 or 2400 mg/day
  Interventions: Drug: GSK1838262
- GSK 1838262 3000 mg/day (Active Comparator): 600 or 1200 or 1800 or 2400 or 3000 mg/day
  Interventions: Drug: GSK1838262

INTERVENTIONS:
Drug: GSK1838262 — Flexible dosing: 1200 mg/day, 1800 mg/day, 2400 mg/day and 3000 mg/day
  Other Names: XP13512
  Arms: GSK 1838262 1200 mg/day; GSK 1838262 1800 mg/day; GSK 1838262 2400 mg/day; GSK 1838262 3000 mg/day
Drug: Placebo — Placebo-control
  Arms: Placebo

SUMMARY:
Purpose of the study is to evaluate dose response relationship, efficacy, safety and tolerability of target doses of GSK1838262 compared to placebo in the prophylactic treatment of migraine headache. Once subjects complete the baseline and meet the randomization criteria, they will complete a 5-wk flexible titration period and then enter the 12 week maintenance period.

DETAILED DESCRIPTION:
MPX111381 is a multicenter, randomized, double-blind, placebo-controlled, parallel group, flexible-dose evaluation of GSK1838262 1200 mg/day, 1800 mg/day, 2400 mg/day and 3000 mg/day compared with placebo in the prophylactic treatment of migraine headache.

Subjects 18 years of age must have experienced at least three migraine headache attacks (with or without aura according to 2004 International Headache Society [IHS] criteria 1.1 and 1.2.1) per month during the 3 months prior to screening and at least four migraine headache days but less than 15 total headache days (migraine or non-migraine) per month during the 3 months prior to screening and must maintain this requirement throughout the last 4 weeks of the baseline period. Approximately 528 subjects from approximately 53 centers in North America will be randomized in a 2:1:2:2:1 ratio to the following treatment groups: placebo, GSK1838262 1200 mg/day, 1800 mg/day, 2400 mg/day and 3000 mg/day. Investigational product will be administered twice daily (morning and evening) with food (e.g., meal or snack).

The study will consist of six study periods for a total study duration of up to 30 weeks: Screening (2 weeks), baseline (including randomization, 6 weeks), flexible titration (5 weeks), maintenance (12 weeks), taper (3 weeks) and post-treatment (2 weeks). The flexible titration administration of investigational product is designed to allow subjects to reach the target dose for maintenance treatment or, if unable to reach this target dose, to achieve a maximum tolerated dose for maintenance treatment. Subjects will have the opportunity to undergo a single dose (600 mg/day) downward adjustment during the flexible titration period if intolerability at the current dose occurs. Subsequently, if a single dose downward adjustment has occurred, no further dose adjustments in the study (upward or downward) will be permitted.

ELIGIBILITY:
Inclusion criteria:

* Outpatient subjects aged 18 years or older.
* Females of non-childbearing potential. If of child-bearing potential, is not lactating and has a negative pregnancy test 7 days prior to study treatment initiation and agrees to use one of the GlaxoSmithKline (GSK)-specified highly effective methods for avoiding pregnancy.
* Subjects suffering from migraine headache with or without aura, according to 2004 IHS criteria 1.1 and 1.2.1.
* Subject has had a history of migraine headache for at least one year, and the age of onset was prior to 50 years.
* Subject has consistent migraine headache over time (i.e., incidence and severity).
* Subject has had at least three migraine headache attacks per month during the 3 months prior to screening and maintains this requirement during the last 4 weeks of the baseline period
* Subject has had at least four migraine headache days but less than 15 total headache days (migraine or non-migraine) per month during the 3 months prior to screening and maintains this requirement during the last 4 weeks of the baseline period.
* Subject is able to distinguish migraine headache attacks as discrete from other headaches (i.e., tension-type headaches).
* Subject has the ability to read, comprehend and legibly and reliably record information in paper and electronic format as required by the protocol.
* Subject must be able to provide written informed consent prior to participation in the study. The contents and process of obtaining informed consent will be in accordance with all applicable regulatory requirements.

Exclusion Criteria:

* Subject has a history of ergotamine, triptan, opioid, and/or combination pain medication use on >/=10 days per month on a regular basis for >/= 3 months.
* Subject has failed more than 2 adequate treatments of migraine prophylaxis -where failure is defined as a lack of efficacy with treatment duration of at least 8 weeks.
* Subject has history of simple analgesic use on >/=15 days per month for >/=3months.
* Subject is unable to discontinue prohibited medications during the 2-week screening period and throughout the duration of the study including beta-blockers, benzodiazepines, tricyclic antidepressants, calcium channel blockers, antiepileptic drugs, bupropion or serotonergic noradrenergic reuptake inhibitors (SNRIs).
* Subjects who have taken gabapentin or pregabalin previously for the prophylactic treatment of migraine headache. Subjects who have taken gabapentin or pregabalin for treatment of conditions other than migraine are eligible provided, (1) their total exposure to gabapentin and pregabalin is less than 3 months during the preceding 12 months, and (2) the subject stopped taking gabapentin or pregabalin for at least 3 months prior to baseline.
* Subject has a history of cluster headaches or basilar, ophthalmoplegic, hemiplegic, or transformed migraine headaches.
* Subject has a current or past history of seizure disorder.
* Subject has any of the following medical conditions, laboratory abnormalities or disorders:
* Hepatic impairment defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2x upper limit of normal (ULN) or alkaline phosphatase or bilirubin >1.5x ULN
* Chronic hepatitis B or C with a positive Hepatitis B surface antigen (HBsAg) or Hepatitis C Core Antigen Antibody (Hep C antibody)
* Impaired renal function defined as either creatinine clearance <60 mL/min (estimation of creatinine clearance by Cockroft and Gault Method) or renal dysfunction requiring hemodialysis
* Corrected QT (QTc) interval >/= 450 msec based on the average QTc value of triplicate electrocardiograms (ECGs) obtained by the central ECG reader over a brief recording period
* QTc interval >/= 480 msec for subjects with Bundle Branch Block based on the average QTc value of triplicate ECGs obtained by the central ECG reader over a brief recording period
* Uncontrolled hypertension at screen or at time of randomization (sitting systolic blood pressure [SBP] >160 mmHg and/or sitting diastolic blood pressure [DBP] >90 mmHg)
* Medical condition or disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of GSK1838262, or, in the investigator's judgement:
* Is considered to be clinically significant and may pose a safety concern, or,
* Could interfere with the accurate assessment of safety or efficacy, or,
* Could potentially affect a subject's safety or study outcome.
* Subject meets criteria as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) for a major depressive episode or for active significant psychiatric disorders within the past year, including dementia, general anxiety disorder, psychotic disorders or bipolar disorder.
* Subjects with a history of depression that is in remission, with or without antidepressant treatment, may participate, unless a stable antidepressant regimen includes a prohibited medication.
* Antidepressant medication may not be changed or discontinued to meet entry criteria and must be stable for at least 3 months prior to screening.
* Subject has a history of clinically significant drug or alcohol abuse as defined by DSM IV TR or is unable to refrain from substance abuse throughout the study.
* Subject is currently participating in another clinical study in which the subject is, or will be exposed to an investigational or non-investigational drug or device.
* Subject has participated in a clinical study in which the subject was exposed to an investigational or non investigational drug or device:
* Within the preceding month for studies unrelated to the current illness (migraine headaches), or
* Within the preceding 3 months for studies related to the current illness (migraine headaches).
* Subjects who have taken botulinum toxin type A (Botox) within the past 6 months.
* Subject has a history of an allergic reaction, or a medically significant adverse reaction to the investigational product or excipients, which, in the opinion of the investigator, makes a subject unsuitable for participation in the study.
* Subject is felt to be at risk of non-compliance (e.g., for taking investigational product or for completing the electronic diary [e-diary]), in the investigator's opinion.
* Subject is a pregnant or nursing woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (51):
- United States (40):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Redlands, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Westlake Village, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Sunrise, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Golden Valley, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, West Chester, Ohio
  - GSK Investigational Site, Westerville, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Canada (11):
  - GSK Investigational Site, Penticton, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

REFERENCES:
- [Derived] Silberstein S, Goode-Sellers S, Twomey C, Saiers J, Ascher J. Randomized, double-blind, placebo-controlled, phase II trial of gabapentin enacarbil for migraine prophylaxis. Cephalalgia. 2013 Jan;33(2):101-11. doi: 10.1177/0333102412466968. Epub 2012 Nov 19. PMID 23165696

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 3 subjects who were randomized but did not take investigational product, and, therefore, were not included in the Safety, Intent to Treat (ITT), or Per Protocol (PP) population.
Groups:
- Placebo: Oral GEn (XP13512) placebo
- GEn 1200 mg: Oral gabapentin enacarbil (GEn; XP13512/GSK1838262). Week 1: 600 mg/day. Weeks 2-17: 1200 mg/day.
- GEn 1800 mg: Oral gabapentin enacarbil (GEn; XP13512/GSK1838262). Week 1: 600 mg/day. Week 2: 1200 mg/day. Weeks 3-17: 1800 mg/day
- GEn 2400 mg: Oral gabapentin enacarbil (GEn; XP13512/GSK1838262). Week 1: 600 mg/day. Week 2: 1200 mg/day. Week 3: 1800 mg/day. Weeks 4-17: 2400 mg/day
- GEn 3000 mg: Oral gabapentin enacarbil (GEn; XP13512/GSK1838262). Week 1: 600 mg/day. Week 2: 1200 mg/day. Week 3: 1800 mg/day. Weeks 4: 2400 mg/day. Weeks 5-17: 3000 mg/day.
Period: Overall Study
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Started | 129 | 67 | 134 | 134 | 62
Completed | 95 | 49 | 88 | 97 | 37
Not Completed | 34 | 18 | 46 | 37 | 25
Not completed — Adverse Event | 11 | 4 | 17 | 16 | 13
Not completed — Participant Withdrew Consent | 8 | 4 | 14 | 7 | 4
Not completed — Protocol Violation | 6 | 5 | 4 | 5 | 3
Not completed — Lost to Follow-up | 3 | 4 | 5 | 5 | 3
Not completed — Lack of Efficacy | 6 | 1 | 1 | 3 | 1
Not completed — Investigator Discretion | 0 | 0 | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat population
Groups:
- Placebo: Oral GEn (XP13512) placebo on Weeks 1-17
- Total: Total of all reporting groups
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg | Total
Number analyzed (Participants) | 128 | 66 | 134 | 133 | 62 | 523
Age Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.72) | 39.4 (9.74) | 37.7 (11.75) | 39.0 (12.04) | 39.1 (11.78) | 39.2 (11.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 52 | 115 | 105 | 46 | 429
  Male | 17 | 14 | 19 | 28 | 16 | 94
Race/Ethnicity, Customized [Number; unit: participants]
  White | 108 | 54 | 107 | 112 | 53 | 434
  African American/African Heritage (AA) | 11 | 8 | 15 | 11 | 6 | 51
  American Indian (AI) or Alaska Native (AN) | 2 | 1 | 3 | 1 | 0 | 7
  Asian | 4 | 3 | 6 | 6 | 3 | 22
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  AA/African Heritage and AI or AN and White | 0 | 0 | 0 | 1 | 0 | 1
  AA/African Heritage and White | 0 | 0 | 2 | 1 | 0 | 3
  AI or AN and White | 1 | 0 | 1 | 0 | 0 | 2
  Asian and White | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in the Number of Migraine Headache Days (MHD) During the Last 4 Weeks of Treatment Prior to Taper
Description: A migraine headache day is defined as a calendar day with any occurrence of migraine headache pain of at least 30 minutes in duration. Change from baseline was calculated as the mean number of MHD over the last 4 weeks of treatment prior to taper minus the number at baseline using the Last Observation Carried Forward (LOCF). The last 4-week treatment phase is based on the last 4 weeks prior to taper for each participant.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: Intent to treat (ITT). There were 3 subjects who were randomized but did not take investigational product, and, therefore were not included in the Safety, ITT, or Per Protocol (PP) population.
Measure: Least Squares Mean (Standard Error); unit: Migraine Headache Days (MHD)
Groups:
- Average of GEn 1800/2400 mg: Average of GEn 1800 mg group and GEn 2400 mg group
Arm/Group | Placebo | Average of GEn 1800/2400 mg | GEn 1800 mg | GEn 2400 mg
Number analyzed (Participants) | 128 | 261 | 131 | 130
Migraine Headache Days (MHD) | -3.8 (0.38) | -3.6 (0.26) | -3.8 (0.37) | -3.3 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Average of GEn 1800/2400 mg; Test type: Superiority or Other; p = 0.579, ANCOVA — A combination of a sequential method and the Hochberg procedure has been used to maintain the overall experiment-size alphas level of 0.05 for the comparison of GEn vs. placebo; An ANCOVA model with baseline number of MHD and IHS Headache Classification for presence or absence of aura as covariates was used; Adjusted mean difference versus placebo = 0.3, 95% CI 2-sided [-0.6 to 1.1] — Adjusted mean difference versus placebo

2. Secondary Outcome: Mean Change From Baseline in the Number of MHD in All Study Phases
Description: A migraine headache day is defined as a calendar day with any occurrence of migraine headache pain of at least 30 minutes in duration. Change from baseline and the last 4 weeks of treatment prior to taper were calculated means of the number of migraine headache days using the Last Observation Carried Forward (LOCF). Change from baseline is calculated as post-baseline minus baseline. The last 4-week treatment phase is based on the last 4 weeks prior to taper for each participant.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Migraine Headache Days (MHD)
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 124 | 59 | 119 | 124 | 59
Migraine Headache Days (MHD)
  Baseline to Titration(n=124, 59, 119, 124, 59) | -2.434 (0.3621) | -1.920 (0.5224) | -2.431 (0.3375) | -2.573 (0.3352) | -2.325 (0.5055)
  Baseline to 2nd 4-Week (n=124, 59, 119, 124, 59) | -3.595 (0.3784) | -2.739 (0.6897) | -3.953 (0.3794) | -3.360 (0.4201) | -3.520 (0.5669)
  Baseline to 3rd 4-Week (n=124, 59, 119, 124, 59) | -3.865 (0.3992) | -3.171 (0.6660) | -3.9888 (0.3810) | -3.439 (0.4483) | -3.220 (0.6594)
  Baseline to Maint Phase (n=112, 54, 101, 107) | -3.846 (0.3589) | -2.854 (0.6565) | -4.047 (0.3368) | -3.794 (0.3761) | -3.723 (0.6492)
  Baseline to Treat Phase (n=118, 56, 113, 118, 56) | -3.396 (0.3422) | -2.834 (0.5640) | -3.579 (0.3140) | -3.393 (0.3388) | -3.193 (0.5165)
  Baseline to 1st 4-Week (n=124, 59, 119,124, 59) | -3.147 (0.4043) | -2.191 (0.6758) | -3.424 (0.3204) | -3.419 (0.3941) | -2.974 (0.5522)

3. Secondary Outcome: Adjusted Mean Change From Baseline in the Number of Migraine Attacks
Description: A migraine attack is defined as a migraine headache of at least 30 minutes in duration and may also include recurring non-migraine or migraine headaches . Change from baseline and the last 4 weeks of treatment prior to taper were calculated means of the number of migraine attacks using the Last Observation Carried Forward (LOCF). The last 4-week treatment phase is based on the last 4 weeks prior to taper for each participant.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Migraine Attacks
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 59 | 114 | 123 | 58
Migraine Attacks | -2.2 (0.15) | -2.2 (0.22) | -2.3 (0.16) | -2.1 (0.15) | -2.6 (0.22)

4. Secondary Outcome: Mean Change From Baseline in the Number of Migraine Headache Periods (MHP)
Description: A migraine headache period is a 24-hour block of time that begins at the onset of a migraine event . The 24-hour period is not linked directly with a calendar day. The change from baseline and the last 4 weeks of treatment prior to taper were calculated means of the number of migraine headache periods using the Last Observation Carried Forward (LOCF). The last 4-week treatment phase is based on the last 4 weeks prior to taper for each participant.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Migraine Headache Periods (MHP)
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 59 | 114 | 123 | 58
Migraine Headache Periods (MHP) | -3.3 (0.35) | -3.0 (0.50) | -3.6 (0.36) | -3.0 (0.34) | -3.2 (0.50)

5. Secondary Outcome: Change From Baseline in the Mean Migraine Attack Duration
Description: The total duration of a migraine attack is measured from migraine attack onset until the resolution of the attack measured in hours and may include more than 1 headache event. The duration is assessed using a Daily Migraine Diary. Change from baseline and the last 4 weeks of treatment prior to taper were calculated means of the number of migraine headache days using the Last Observation Carried Forward (LOCF). Change from baseline is calculated as post-baseline minus baseline. The last 4-week treatment phase is based on the last 4 weeks prior to taper for each participant.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 99 | 52 | 89 | 102 | 44
Hours | -0.97 (3.355) | 3.01 (5.720) | -2.93 (3.658) | 2.59 (5.000) | 9.82 (9.975)

6. Secondary Outcome: Change From Baseline in the Mean Peak Migraine Pain Severity
Description: Peak Migraine Pain Severity was measured using a 4-point scale (0=none, 1=mild, 2=moderate, or 3=severe) on a participant self assessed Daily Migraine Diary. The scale measured the maximum pain severity across all headache events considered to be one attack.. Change from baseline and the last 4 weeks of treatment prior to taper were calculated means of the number of migraine headache days using the Last Observation Carried Forward (LOCF). The last 4-week treatment phase is based on the last 4 weeks prior to taper for each participant.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 99 | 52 | 89 | 102 | 62
Scores on a Scale | -0.12 (0.058) | -0.13 (0.086) | -0.12 (0.055) | -0.04 (0.050) | -0.09 (0.080)

7. Secondary Outcome: Mean Change From Baseline to the Last 4-Week Treatment Phase in the Number of Days of Acute Migraine Medication Use
Description: The Number of Days of Acute Migraine Medication Use was assessed via the participant-assessed Daily Migraine Diary.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 59 | 114 | 123 | 58
Days | -2.0 (0.28) | -2.3 (0.39) | -2.7 (0.28) | -2.2 (0.27) | -2.1 (0.40)

8. Secondary Outcome: Mean Change From Baseline to the Last 4-Week Treatment Phase in the Number of Acute Migraine Medication Doses Administered
Description: The Number of Acute Migraine Medication Doses Administered was captured via the participant-assessed Daily Migraine Diary.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Acute Medication Doses Admin.
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 59 | 114 | 123 | 58
Acute Medication Doses Admin. | -4.5 (0.69) | -4.8 (0.97) | -5.8 (0.70) | -5.1 (0.67) | -4.5 (0.69)

9. Secondary Outcome: Mean Change From Baseline to the Last 4-Week Treatment Phase in the Number of Acute Migraine Medication Doses Administered by Triptan Use
Description: The Number of Acute Migraine Medication Administered was measured via the participant-assessed Daily Migraine Diary.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Acute Migraine Medication Dose
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 59 | 114 | 123 | 58
Acute Migraine Medication Dose
  Triptan Use (n= 72, 30, 65, 63, 32) | -3.3 (0.88) | -2.9 (1.35) | -4.9 (0.91) | -4.3 (0.93) | -2.6 (1.31)
  Not a Triptan User (n = 48, 29, 49, 60, 26) | -6.3 (1.06) | -6.7 (1.36) | -6.9 (1.05) | -6.0 (0.95) | -6.8 (1.44)

10. Secondary Outcome: Mean Change From Baseline to the Last 4-Week Treatment Phase in the Number of Acute Migraine Medication Doses Administered by Opioid Use
Description: The Number of Acute Migraine Medication Doses Administered by Opioid Use was measured via the participant-assessed Daily Migraine Diary.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 59 | 114 | 123 | 58
Days
  Opioid Use (n=20, 7, 14, 26, 10) | -1.7 (1.66) | 1.4 (2.81) | -3.2 (1.97) | -6.0 (1.45) | -5.1 (2.34)
  Non-Opioid Use (n=100, 52, 100, 97, 48) | -5.1 (0.75) | -5.7 (0.75) | -6.2 (0.74) | -4.9 (0.75) | -4.4 (1.08)

11. Secondary Outcome: Mean Change From Baseline to the Last 4-Week Treatment Phase in the Number of Acute Migraine Medication Doses Administered by Prescription Headache Medication Use
Description: The Number of Acute Migraine Medication Doses Administered by Prescription Headache Medication use was measured via the participant-assessed Daily Migraine Diary.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Acute Migraine Medication Doses
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 59 | 114 | 123 | 58
Acute Migraine Medication Doses
  Uses Prescription HA meds (n=89, 38, 80, 88, 39) | -3.6 (0.78) | -3.5 (1.19) | -4.9 (0.82) | -4.0 (0.78) | -3.3 (1.18)
  Uses OTC HA meds only (n=31, 21, 34, 35, 19) | -6.9 (1.31) | -7.2 (1.59) | -7.8 (1.25) | -7.9 (1.23) | -6.9 (1.68)

12. Secondary Outcome: Mean Change From Baseline in Percentage of Migraine Attacks With Each of the Following Migraine Symptoms: Aura, Nausea, Vomiting, Photophobia, Phonophobia
Description: The endpoint is defined as the percentage of attacks with each symptom (separately) for each study phase. Migraine symptoms aura, nausea, vomiting, photophobia, and phonophobia are defined as the presence of each migraine symptom during any of the headache events within an attack.
Time Frame: Baseline and last 4 weeks of treatment prior to taper (up to Week 17)
Population: ITT Population
Measure: Mean (Standard Error); unit: Percentage of MA with migraine symptoms
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 125 | 62 | 123 | 121 | 59
Percentage of MA with migraine symptoms
  Aura (n=99, 52, 89, 102, 44) | -7.4 (3.640) | -3.37 (4.834) | -7.43 (3.230) | -0.72 (3.044) | 1.21 (4.372)
  Nausea (n=125, 62, 123, 121, 59) | -7.8 (2.73) | -3.6 (3.92) | -8.4 (3.01) | -5.4 (2.50) | 1.4 (3.31)
  Vomiting (n=99, 52, 89, 102, 44) | 0 (2.60) | -0.9 (2.98) | -0.4 (3.01) | 3.7 (0.4) | 0.4 (4.83)
  Photophobia (n=99, 52, 89, 102, 44) | -1.9 (2.82) | -3.5 (4.09) | -2.1 (2.86) | -5.5 (2.64) | 0.1 (2.49)
  Phonophobia (n=99, 52, 89, 102, 44) | -5.4 (3.14) | 1.2 (3.05) | -0.7 (3.42) | -7.4 (2.88) | 3.6 (1.93)

13. Secondary Outcome: Percentage of Participants Classified as Responders for Each of the Following Measures: Migraine Headache Days, Migraine Attacks, and Migraine Headache Periods
Description: A responder is defined as a participant who achieved at least a 50% reduction from baseline for the indicated measures.
Time Frame: Baseline to the Last 4 weeks of treatment
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 65 | 31 | 70 | 69 | 40
percentage of participants
  Migraine headache days (n=65, 26, 68, 67, 38) | 54 | 44 | 60 | 54 | 66
  Migraine attacks (n=64, 31, 67, 67, 39) | 53 | 53 | 59 | 54 | 67
  Migraine headache periods (n=65, 27, 70, 69, 40) | 54 | 46 | 61 | 56 | 69

14. Secondary Outcome: Number of Participants Who Were "Much Improved" or "Very Much Improved" on the 7-point Likert Patient Global Impression of Change (PGIC) Scale Using LOCF at Week 17
Description: The PGIC is a single question measured on the 7-point Likert Scale (1 = "very much improved"; 2 = "much improved"; 7 = "very much worse"). A responder is defined as being "very much improved" or "much improved."
Time Frame: Week 17
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 123 | 57 | 115 | 121 | 55
participants | 71 | 40 | 84 | 81 | 36

15. Secondary Outcome: Number of Participants Who Were "Much Improved" or "Very Much Improved" (Responders) on the 7-point Likert Clinical Global Impression of Change (CGIC) Scale Using LOCF at Week 17
Description: The CGIC is a single question measured on a 7-point Likert Scale. (1 = "very much improved"; 2= "much improved, and 7 = "very much worse") designed to give an assessment of treatment from a clinician's perspective. A responder is defined as being 'Very much improved' or 'much improved'.
Time Frame: Week 17
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 124 | 57 | 116 | 120 | 55
Participants | 75 | 40 | 84 | 85 | 32

16. Other Pre Specified Outcome: Mean Change From Baseline in Migraine Specific Quality of Life Questionnaire (MSQ v2.1) Composite Score and Subscales (Role Function Restrictive, Role Function, Preventive, & Emotional Function) at Week 17
Description: The MSQ is a 14-item health-related quality of life (HRQOL) questionnaire. Participants provide responses using a 6-point Likert scale (1=None of the time, 2= A little bit of the time, 3=Some of the time, 4=A good bit of the time, 5=Most of the time, 6=All of the time) that are then recoded with a final item value where 1=6, 2=5, 3=4, 4=3, 5=2, and 6=1. The scale measures 3 independently scored dimensions (Role Function Restrictive, Role Function, Preventive, and Emotional Function) of HRQOL that are affected by migraine. For each dimension, a higher score indicates a better health status.
Time Frame: Baseline and Week 17
Population: ITT Population
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 57 | 115 | 121 | 62
units on a scale
  Role Function Restrictive | 30.7 (2.31) | 38.7 (3.12) | 37.1 (2.38) | 32.8 (2.28) | 30.9 (3.73)
  Role Function Preventive | 22.7 (1.98) | 28.6 (2.67) | 28.0 (2.04) | 23.9 (1.96) | 22.4 (3.20)
  Emotional Function | 29.7 (2.56) | 37.0 (3.46) | 34.8 (2.64) | 30.4 (2.54) | 25.7 (4.14)

17. Other Pre Specified Outcome: Mean Change From Baseline in the Headache Impact Test (HIT-6) Total Scores at Week 17
Description: The HIT is a 6-item, self-administered HRQOL questionnaire used to measure six areas that impact headaches have on participants' ability to function on the job, at school, at home, and in social situations. Participants provide responses to questions using a 5-point Likert-type scale. All item values range from 6 to13.The total scores range from 36 to 78, where higher scores indicate greater impact on a participant's life.
Time Frame: Week 17
Population: ITT Population
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 120 | 57 | 115 | 121 | 54
Points on a scale | -10.0 (0.95) | -12.2 (1.28) | -11.8 (0.98) | -9.8 (0.94) | -10.3 (1.53)

18. Other Pre Specified Outcome: Mean Change From Baseline in Productivity as Measured by Lost Time Equivalents (LTE) - (Work Activities, Non-work Activities, and Combination of Work and Non-work Activities)
Description: Productivity, as measured by LTE, is a metric used to assess productivity loss in migraine. It is a composite measure of presenteeism (continued to work while under the influence of migraine symptoms) and absenteeism (time missed from work due to migraine), and can be applied to productivity for work and non-work activities. Productivity data were collected via an e-diary, and productivity measures were summarized for each study phase by averaging each measure across migraine attacks for each participant.
Time Frame: Week 17
Population: ITT Population
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 99 | 52 | 89 | 102 | 44
Hours
  Lost Work Time (n=52, 23, 41, 35, 17) | -0.8 (0.49) | -0.3 (0.73) | -0.9 (0.55) | -0.1 (0.59) | 0.8 (0.85)
  Lost Activity Time (n=99,52, 89, 102, 44) | 0.1 (0.74) | -0.1 (1.02) | -1.2 (0.78) | -1.0 (0.73) | 1.7 (1.11)
  Lost Time Equivalents (n=99, 52, 89, 102, 44) | -0.2 (0.83) | -0.5 (1.14) | -1.7 (0.87) | -1.1 (0.082) | 2.1 (1.24)

19. Other Pre Specified Outcome: Assessment of Treatment Satisfaction Using the Patient Perception of Migraine Questionnaire (PPMQ-R) at Week 17
Description: Three global treatment satisfaction items from the PPMQ included satisfaction or dissatisfaction with Medication Effectiveness, Medication Side Effects, and Overall Medication. Each item on the PPMQ uses a 7-point satisfaction scale (1 = Very Satisfied to 7 = Very Dissatisfied). Satisfied participants include those reporting "Very Satisfied" (scale value = 1) or "Satisfied" (scale value = 2) on the scale.
Time Frame: Week 17
Population: ITT Population
Measure: Number; unit: Percentage of Patients
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Number analyzed (Participants) | 123 | 57 | 118 | 120 | 54
Percentage of Patients
  How Effective Overall | 74 | 39 | 84 | 81 | 36
  Side Effects of the Medication | 79 | 32 | 72 | 75 | 28
  Overall Satisfaction with Medication | 76 | 39 | 84 | 84 | 34

ADVERSE EVENTS:
Description: Serious adverse events (AEs) and non-serious AEs were collected in the Safety Population, comprised of all randomized participants who took at least one tablet of investigational product. There were no participants who took drug and did not have at least one post-baseline efficacy assessment; thus, the Safety and ITT Populations are the same.
Arm/Group | Placebo | GEn 1200 mg | GEn 1800 mg | GEn 2400 mg | GEn 3000 mg
Serious Adverse Events (participants affected / at risk) | 2/128 | 0/66 | 2/134 | 1/133 | 4/62
Other Adverse Events (participants affected / at risk) | 86/128 | 44/66 | 99/134 | 101/133 | 47/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=128) | GEn 1200 mg (N=66) | GEn 1800 mg (N=134) | GEn 2400 mg (N=133) | GEn 3000 mg (N=62)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choleslithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=128) | GEn 1200 mg (N=66) | GEn 1800 mg (N=134) | GEn 2400 mg (N=133) | GEn 3000 mg (N=62)
Dizziness (Nervous system disorders) | 8 | 16 | 43 | 35 | 11
Fatigue (General disorders) | 9 | 10 | 12 | 14 | 3
Nausea (Gastrointestinal disorders) | 12 | 3 | 15 | 12 | 6
Somnolence (Nervous system disorders) | 6 | 6 | 7 | 14 | 9
Weight increased (Investigations) | 7 | 4 | 8 | 9 | 4
Upper respiratory track infection (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 4 | 9 | 5
Constipation (Gastrointestinal disorders) | 3 | 4 | 7 | 8 | 5
Dry mouth (Skin and subcutaneous tissue disorders) | 3 | 4 | 6 | 5 | 3
Nasopharyngitis (Infections and infestations) | 8 | 3 | 4 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 1 (1) | 1 (1) | 7 | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 | 1 (1) | 3 | 7 | 2
Influenza (Infections and infestations) | 4 | 1 (1) | 3 | 4 | 3
Insomnia (Psychiatric disorders) | 1 (1) | 4 | 1 (1) | 6 | 2
Oedema (General disorders) | 4 | 4 | 1 (1) | 3 | 2
Sinusitis (Infections and infestations) | 3 | 4 | 3 | 3 | 1 (1)
Balance (Nervous system disorders) | 1 (1) | 2 | 2 | 6 | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 | 2 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 6 | 1 (1) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.